CLINICAL TRIAL: NCT01105702
Title: Temozolomide, Bevacizumab, Lithium and Radiation Treatment for Newly Diagnosed High Grade Glioma: A Phase II Study
Brief Title: Temodar (Temozolomide), Bevacizumab, Lithium and Radiation for High Grade Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry); Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 07-712
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Brain Cancer
Keywords: brain tumor; brain cancer; glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Temozolomide; Bevacizumab; Lithium Carbonate; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TBL/RT (Experimental): Cycle 1(One 42-day cycle)
  * Temozolomide 75 mg/m^2 orally (42 consecutive days), beginning the night prior to the first radiation treatment
  * Radiation within 3-5 weeks of surgery
  * Bevacizumab 10mg/kg, IV, starting 29 (+3) days post surgery and every 2 weeks
  Treatment Cycles 2-7 (28 days per cycle)
  * Temozolomide at a dose of 150 mg/m^2 on Days 1-7
  * Bevacizumab 10 mg/kg on Day 8 and Day 22
  * Initiate Lithium carbonate treatment at 300 mg, orally, twice a day; dose increased every 7 days up to 600mg, orally, twice a day, to a serum lithium level of 0.8-1.2 mEq/L.
  Interventions: Drug: Temozolomide; Drug: Bevacizumab; Drug: Lithium Carbonate; Radiation: Radiation

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodar
Drug: Bevacizumab
  Other Names: Avastin
Drug: Lithium Carbonate
  Other Names: Lithobid
Radiation: Radiation

SUMMARY:
This pilot phase II trial studies how well giving temozolomide, bevacizumab, lithium carbonate, and radiation therapy works in treating patients with newly diagnosed high grade glioma.

DETAILED DESCRIPTION:
Treatment of high grade glioma (HGG) with anti-angiogenic therapy results in clinical improvement and prolonged progression-free survival (PFS). However, mant patients experience diffuse recurrence and treatment failure. This is a phase II trial testing the feasibility of adding lithium carbonate, previously shown to have anti-invasive properties in HGG, to bevacizumab and chemoradiation following surgical resection of HGG.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed high grade glioma (WHO Grade III and IV)
* Brain magnetic resonance imaging (MRI) scan with gadolinium contrast
* Patient must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >= 1,500/mm^3;
  * Platelet count >=100,000/mm^3;
  * Hemoglobin >= 10g/dL;
  * Blood urea nitrogen and serum creatinine both =< 1.5 times upper limit of normal (ULN);
  * Total bilirubin both =< 1.5 times ULN;
  * SGOT and SGPT both =< 3 times ULN;
  * Alkaline phosphatase =< 2 times ULN.
* >=18 years of age;
* Karnofsky Performance Score >= 70;
* Life expectancy >= 8 weeks;
* Negative serum or urine beta-hCG pregnancy test at screening for patients of child bearing potential;
* Men and women with reproductive potential must agree to use an acceptable method of birth control (surgical, hormonal or double barrier, ie, condom and diaphragm) during treatment and for 6 months after completion of treatment;
* Patient or their legal proxy must provide written informed consent prior to registration on study;
* Residual measurable disease.

Exclusion Criteria:

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study;
* Prior radiation therapy to the brain;
* Prior treatment with Chemotherapy or Targeted agent
* Previous (within last 5 years) or current malignancies at other sites except for adequately treated basal cell or squamous cell skin cancer in situ carcinoma of the cervix;
* (Uncontrolled High blood pressure >150/100
* Common Terminology Criteria Adverse Event 3.0 >= Grade 2 congestive heart failure (CHF);
* History of myocardial infarction within 6 months;
* History of stroke within 6 months;
* Clinically significant peripheral vascular disease;
* Evidence of bleeding diathesis or coagulopathy;
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of bevacizumab or anticipation of need for major surgical procedure during the course of the study;
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to study enrollment;
* Urine protein/Creatinine ratio >= 2.0 at screening;
* Serious, non-healing wound, ulcer, or bone fracture;
* Inability to comply with study and/or follow-up procedures;
* Glioma showing active intratumoral bleeding;
* Patients on enzyme-inducing anti-epileptic drugs;
* Known Positive HIV-1, hepatitis B surface antigen, or hepatitis C antibody;
* Medications like nonsteroidal antiinflammatory drugs, antipsychotics, iodides, and angiotensin-converting enzyme inhibitor, If they are receiving them, they must have been discontinued for 7 days prior to initiating lithium;
* Any previous cytotoxic drug therapies, excluding corticosteroids and temozolomide concurrent with radiation therapy;
* Any known genetic cancer-susceptibility syndromes;
* Acute infection: any active viral, bacterial, or fungal infection that requires specific therapy.
* Active uncontrolled infection - examples include sexually transmitted disease, herpes, scrofula, malaria, etc.;
* Fever > 101.5 degrees Fahrenheit;
* Unstable or severe intercurrent medical conditions such as unstable angina, uncontrolled arrythmias, Crohn's disease, ulcerative colitis, psoriasis, etc.;
* Implantation of Gliadel wafers at surgery;
* Patients with organ allografts; and
* Allergies to reagents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gruber, MD, Principal Investigator — New York University Cancer Institute
Locations (2):
- United States (2):
  - Overlook Hospital, Summit, New Jersey
  - New York University Clinical Cancer Center, New York, New York

REFERENCES:
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2010 to June 2012, 28 patients were enrolled from New York University Langone Medical Center and Outlook Hospital, Summit, NJ.
Period: Overall Study
Arm/Group | TBL/RT
Started | 28
Completed | 10
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: All patients enrolled
Arm/Group | TBL/RT
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 26
  Asian | 1
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
World Health Organization Grade (staging) [Number; unit: participants] — Grade III: Malignant although there is not always a big difference between grade II and grade III tumors. The cells of a grade III tumor are actively reproducing abnormal cells, which grow into nearby normal brain tissue. These tumors tend to recur, often as a grade IV.
  Grade IV: These are the most malignant tumors. They reproduce rapidly, can have a bizarre appearance when viewed under the microscope, and easily grow into nearby normal brain tissue. These tumors form new blood vessels so they can maintain their rapid growth.
  participants
    Grade III | 8
    Grade IV | 20

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS)
Description: PFS defined as time from date of diagnosis to most recent follow up, disease progression, or death. Disease progress defined as either clinical deterioration or radiographic progressive disease on magnetic resonance imaging (MRI) per updated response assessment in neuro-oncology criteria (Wen, et al).
Time Frame: Up to 50 months
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TBL/RT
Number analyzed (Participants) | 28
months | 9.4 [6.1 to 12.4]

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS defined as time from diagnosis to most recent follow up or death.
Time Frame: Up to 50 months
Population: intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TBL/RT
Number analyzed (Participants) | 28
months | 18.5 [14.7 to 20.8]

3. Secondary Outcome: Number of Patients With Grade 3 or 4 Adverse Events
Description: Adverse events evaluated per CTCAE 3
Time Frame: The whole time while on treatment and 30 days after the treatment
Population: all the patients with treatment
Measure: Number; unit: participants
Groups:
- Grade 3; Grade 4: Cycle 1(One 42-day cycle)
  * Temozolomide 75 mg/m^2 orally (42 consecutive days), beginning the night prior to the first radiation treatment
  * Radiation within 3-5 weeks of surgery
  * Bevacizumab 10mg/kg, IV, starting 29 (+3) days post surgery and every 2 weeks
  Treatment Cycles 2-7 (28 days per cycle)
  * Temozolomide at a dose of 150 mg/m^2 on Days 1-7
  * Bevacizumab 10 mg/kg on Day 8 and Day 22
  * Initiate Lithium carbonate treatment at 300 mg, orally, twice a day; dose increased every 7 days up to 600mg, orally, twice a day, to a serum lithium level of 0.8-1.2 mEq/L.
Arm/Group | Grade 3 | Grade 4
Number analyzed (Participants) | 28 | 28
participants
  Dermatitis | 1 | 0
  DVT | 1 | 0
  Neurologic | 3 | 0
  Pneumonia | 1 | 0
  Rash | 1 | 0
  Cough | 1 | 0
  Hyponatremia | 1 | 0
  Gastrointestinal | 2 | 0
  Febril Neutropenia | 0 | 1
  Neutropenia | 1 | 0
  Thrombocytopenia | 1 | 1
  Somnolence | 1 | 0

ADVERSE EVENTS:
Time Frame: whole time while on treatment plus 30 days after the treatment
Arm/Group | TBL/RT
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TBL/RT (N=28)
Infection with unknown ANC: Wound (Infections and infestations) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
Infection with unknown ANC: Lung (pneumonia) (Infections and infestations) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Infection with unknown ANC: Eye NOS (Infections and infestations) | 1
Pain - Other (Specify, __): jaw (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TBL/RT (N=28)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip): (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 9
Ataxia (incoordination) (Nervous system disorders) | 1
Auditory/Ear - Other (Specify, __): flud in right ear (Ear and labyrinth disorders) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 1
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dental: periodontal disease (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Flushing (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemorrhage, GI: Oral cavity (Gastrointestinal disorders) | 3
Hemorrhage, GI: Rectum (Gastrointestinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory: Nose (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Cardiac disorders) | 1
Infection - Other (Specify, __): thrush (Infections and infestations) | 1
Infection - Other (Specify, __): Urinary tract infection (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Urinary tract NOS (Infections and infestations) | 1
Insomnia (General disorders) | 4
Memory impairment (Nervous system disorders) | 2
Mood alteration: Anxiety (Nervous system disorders) | 3
Mood alteration: Depression (Nervous system disorders) | 2
Mucositis/stomatitis (clinical exam): Stomach (Gastrointestinal disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy): Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Neuropathy: cranial- Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 1
Neuropathy: cranial- sensory facial (Nervous system disorders) | 1
Neuropathy: Cranial-smell (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Nystagmus (Eye disorders) | 1
Pain: Back (Musculoskeletal and connective tissue disorders) | 1
Pain: Bone (Musculoskeletal and connective tissue disorders) | 1
Pain: Chest/thorax NOS (General disorders) | 1
Pain: Dental/teeth/peridontal (Gastrointestinal disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain: Head/headache (Nervous system disorders) | 11
Pain: Middle ear (Ear and labyrinth disorders) | 1
Pain: Stomach (Gastrointestinal disorders) | 1
Platelets (Blood and lymphatic system disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Rash: dermatitis associated with radiation: Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 3
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 1
Sweating (diaphoresis) (General disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 2
Tremor (Nervous system disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Vision-blurred vision (Eye disorders) | 5
Vision-flashing lights/floaters (Eye disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss: (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes